CLINICAL TRIAL: NCT04399226
Title: Efficacy and Safety of Deksmedetomidine-propofol or Ketamine-propofol
Brief Title: Dexmedetomidine-Propofol and Ketamine-Propofol During Upper Gastrointestinal System Sedation
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Assistant Professor, Yuzuncu Yil University
Other Study IDs: umutkan
Record Dates: First submitted 2020-04-29; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia; Reaction
Keywords: Dexmedetomidine, Ketamine, Propofol, Sedation
MeSH Terms: interventions — Dexmedetomidine; Propofol; Ketamine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dexmedetomidine — Group D received 1mg/kg dexmedetomidine+0.5mg/kg propofol intravenous (iv) bolus, 0.5 μg/kg/h dexmedetomidine+ 0.5 mg/kg/h propfol infusion. Group K received 0.125 mL/kg bolus, 0.125 mL/kg/h ketamine+ propofol = ketofol infusion (ketofol was prepared with 4 mg propofol+2 mg ketamine).
  Other Names: propofol; ketamine

SUMMARY:
Sedation with dexmedetomidine-propofol or ketamine-propofol was planned in patients with upper gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Patients between 18 and 60 years in American Society of Anesthesiologists (ASA) I and II groups were included. Patients that had severe organ disease, allergies to study drugs, refused to participate in the study were excluded. Cases were randomized into the dexmedetomidine-propofol group (Group D, n=30) and ketamine-propofol group (Group K, n=30). Cardiac monitoring, peripheral oxygen saturation, bispectral index (BIS) monitoring were performed. Group D received 1mg/kg dexmedetomidine+0.5mg/kg propofol intravenous (iv) bolus, 0.5 μg/kg/h dexmedetomidine+ 0.5 mg/kg/h propfol infusion. Group K received 0.125 mL/kg bolus, 0.125 mL/kg/h ketamine+ propofol = ketofol infusion (ketofol was prepared with 4 mg propofol+2 mg ketamine). Patients were followed up with a Ramsay Sedation Scale (RSS) of≥4. Mean, standard deviation, mean, lowest-highest frequency and ratio values were used in descriptive statistics of the data, SPSS 22.0 program was used for the analyses.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II group
* 60 patients
* between the ages of 18 and 60
* planned to have upper gastrointestinal system (UGIS) endoscopy with sedation,

Exclusion Criteria:

* severe heart, lung, liver disease
* kidney failure,
* bleeding diathesis
* fever,
* infection,
* electrolyte disorder such as hypokalemia, hypocalcaemia, acid-base disorder, hypothermia, allergy to drugs to be used, and study those who refused to be included were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients between 18 and 60 years in American Society of Anesthesiologists (ASA) I and II groups were included. Patients that had severe organ disease, allergies to study drugs, refused to participate in the study were excluded. Cases were randomized into the dexmedetomidine-propofol group (Group D, n=30) and ketamine-propofol group (Group K, n=30).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Demographic data | 2 minutes
  no difference

SECONDARY OUTCOMES:
adverse events | 2 minutes
  Nausea, vomiting and allergic reaction, cough

OTHER OUTCOMES:
sedation depth | 2 minutes
  Measured with BIS

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Esen TEKELİ, MD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
yes